CLINICAL TRIAL: NCT01181362
Title: A Feasibility Study Comparing Head And Neck Endoscopy Procedures In The Upright And Supine Positions
Brief Title: Comparing Head and Neck Endoscopy Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 09-0886-AE
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Comparing Head And Neck Endoscopy in Healthy Patients
Keywords: Endoscopy; Head and Neck region; Scope
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endoscopy (Other)
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Endoscopy — All patients will meet the physician at the Head and Neck centre at PMH, where they will have a topical anesthetic (lidocaine endotracheal aerosol, 10 mg/dose) sprayed into both nostrils. After allowing 5-10 minutes to let the anesthetic take effect, they will have an endoscopy procedure using a flexible scope inserted through the nostrils. The procedure will first be performed while patients are sitting up. During the procedure, patients will be asked to rate their discomfort on a 10-point scale. The endoscope will then be removed. After a short rest (15 minutes), the endoscopy procedure will be repeated with patients lying down. They will again be asked to rate their level of discomfort. After another short rest for recovery, they will meet with the physician to discuss both endoscopic procedures and to complete a questionnaire on discomfort, tolerance and acceptability

SUMMARY:
Intensity Modulated Radiation Therapy planning is based on CT images, with tumour volumes defined on this volumetric information data set. However, target delineation also depends on disease seen endoscopically which may not be visible on CT. We are developing imaging and tracking technology to improve target delineation in Radiation Therapy (RT) planning for head & neck cancer using quantitative registration of 2D endoscopic information with CT data. Diagnostic endoscopy is performed in the upright position. CT images and radiation delivery are obtained with the patient in the supine position. The accuracy of the registration will be improved if performed in the same position to prevent mobile soft tissue structures shifting between the upright and supine positions. Since therapy must be performed in the supine position, we intend to check the feasibility of performing endoscopy in the supine treatment position. We will compare and assess patient comfort and endoscopic sightlines during an endoscopy procedure in both the upright and supine positions.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-70 years of age.
* Willing to give informed consent.

Exclusion Criteria:

* Allergy to topical anesthetic nasal spray (lidocaine).
* Patients who currently have or have had head and neck cancer.
* Currently pregnant or lactating; or serious co-morbid illness (e.g., cardiovascular, pulmonary).
* Psychiatric or addictive disorders which would preclude obtaining informed consent or adherence to protocol.
* Concurrent illness, which prevents the subject from undergoing endoscopy.
* Disorders of the nasal cavity e.g deviated septum

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To compare and assess subject comfort and adequacy of endoscope sightlines during an endoscopy procedure in both the upright and supine positions. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: John Cho, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada